CLINICAL TRIAL: NCT06195202
Title: A Prospective Cohort Study of Serum Estradiol (E2) Levels in Breast Cancer Patients During Endocrine Therapy by High Performance Liquid Chromatography-tandem Mass Spectrometry (LC-MS /MS)
Brief Title: Serum Estradiol (E2) Levels in Breast Cancer Patients During Endocrine Therapy by High Performance Liquid Chromatography-tandem Mass Spectrometry (LC-MS /MS)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cong Xue, Clinical Professor, Sun Yat-sen University
Other Study IDs: B2023-351-01
Record Dates: First submitted 2023-12-24; First posted 2024-01-08 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: LC MS/MS; estradiol
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — serem 1ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AI: Patients with AIs
  Interventions: Drug: AIs
- OFS+AI: Patients with OFS+AIs
  Interventions: Drug: OFS+AIs
- FUL: Patients with FUL
  Interventions: Drug: FUL

INTERVENTIONS:
Drug: AIs — Patients with AIs
  Groups: AI
Drug: OFS+AIs — Patients with OFS+AIs
  Groups: OFS+AI
Drug: FUL — Patients with FUL
  Groups: FUL

SUMMARY:
The investigators intend to conduct a prospective cohort study to detect E2 levels during endocrine therapy in Chinese breast cancer patients using LC-MS/MS methods, and to determine the proportion of patients with premenopausal E2 levels (OFR or E2 insufficiency) during AIs or FUL endocrine therapy. To further explore the correlation between serum E2 levels and the efficacy of endocrine therapy in Chinese patients, so as to ensure the safety and efficacy of endocrine therapy for patients, and pave the way for further providing more accurate individualized treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Histologically confirmed breast cancer;
* Patients with early breast cancer (including natural menopause and artificial menopause using LHRHa), or patients with advanced breast cancer (including natural menopause and artificial menopause using LHRHa) who use AIs (letrozole, anastrozole or exemestane) as adjuvant endocrine therapy, First-line CDK4/6 inhibitors (Palbociclib, Dalpiciclib, Abemaciclib or Ribociclib) +AI endocrine therapy, second-line CDK4/6 inhibitors (Palbociclib, Dalpiciclib, Abemaciclib or Ribociclib) + fluvestrant (FUL) endocrine therapy;
* Patients with needs for hormone testing;
* Standard treatment, complete clinical data, including complete efficacy evaluation and follow-up data.

Exclusion Criteria:

* Breast cancer patients using TAM endocrine therapy;
* In advanced patients, AIs exceeded first-line use (that is, in advanced disease, one endocrine therapy regimen had been used and failed), and FUL exceeded second-line use (that is, more than one endocrine therapy regimen had been used and failed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2023.9-2024.68 Breast cancer patients who received aromatase inhibitor (AIs) or fulvestrant (FUL) endocrine therapy in Sun Yat-sen University Cancer Center and need to test hormone levels.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The serum E2 levels in breast cancer patients during endocrine therapy. | From enrollment to 1 months
  Consistency between 2 methods

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided